CLINICAL TRIAL: NCT01352975
Title: Longitudinal Investigation of Dark Adaptation in Participants With Age-Related Macular Degeneration
Brief Title: Study of Dark Adaptation in Age-Related Macular Degeneration
Status: Active, not recruiting | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110147; 11-EI-0147
Record Dates: First submitted 2011-05-11; First posted 2011-05-12 (Estimated); Last update posted 2025-12-08 (Actual); Status verified 2025-08-20

CONDITIONS: Age-Related Macular Degeneration
Keywords: Dark Adaptation; Age-Related Macular Degeneration (AMD); Natural History; Age Related Macular Degeneration; AMD
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Group 0: participants without AMD (no large drusen or advanced AMD in either eye)
- Group 1: participants with large drusen in study eye and no large drusen or advanced AMD or GA in fellow eye
- Group 2: participants with bilateral large drusen with or without retinal pigment epithelial hypo/hyperpigmentary changes
- Group 3: participants with large drusen in study eye and advanced AMD (CNV and GA) in fellow eye
- Group 4: participants with findings of RPD

SUMMARY:
Background:

* Age-related macular degeneration (AMD) is a leading cause of vision loss in individuals over 55 years of age. It can cause permanent loss of central vision, which is important for seeing fine details and long distances. AMD has two forms: wet AMD and dry AMD. Most people with AMD have dry AMD. But dry AMD can progress to wet AMD. Wet AMD is the more serious form and can result in severe vision loss.
* A method to identify and monitor the early to middle stages of AMD may help researchers develop new treatments to stop the disease before it becomes severe. In early dry AMD, people cannot see well at night. Researchers want to study whether a procedure that measures how the eye adjusts to the dark can help to identify and monitor early to middle dry AMD.

Objectives:

- To evaluate the effectiveness of using a dark adaptation protocol to identify and monitor early to middle dry age-related macular degeneration.

Eligibility:

- People at least 50 years of age who have no AMD. Others who have early to middle dry AMD in at least one eye.

Design:

* People will be screened with a physical examination, medical history, blood and urine tests, and a full eye exam.
* This study will last 5 years and require at least 9 visits to NIH. (First visit; study visits at months 3, 6, 12, 18, and 24; and 3 yearly followup visits).
* Up to 10 people will be asked to come back to the clinic 1 week after their first visit. They will be asked to test the device to be used in the study.
* Participants will have baseline exams. These questions will be about problems that affect their eyes under different lighting conditions.
* At every visit, participants will answer questions about general health and current medications (including any vitamins or supplements). They will also have a full eye exam and a 20- to 40-minute test. This test measures how fast the eyes recover in response to decreasing levels of light. The test also measures how sensitive the eyes are to these conditions.
* Participants will continue to have these tests at the yearly followup examinations. They will be treated with the standard of care for any eye conditions they have or may develop during the study.

DETAILED DESCRIPTION:
Objective: This study is designed to investigate the use of dark adaptation as a functional endpoint for progression of eyes with no to intermediate age-related macular degeneration (AMD). To that aim, correlating structural features (obtained from multimodal imaging) as well as genetic and systemic factors obtained from biospecimens with functional measures (including dark adaptation, visual acuity and low luminance) will be done to understand the relationship of disease relevant factors and to create a model of disease pathogenesis and progression.

Study Population: Two hundred forty (240) participants will be initially accrued; however, up to 280 participants who meet the eligibility criteria may be enrolled. Participants will have varying degrees of severity of AMD (Groups 0, 1, 2, 3 and 4). Group 0 (N=40) is defined as participants without AMD meaning no large drusen (>= 125 microns) or advanced AMD in either eye. Group 1 (N=40) is defined as participants with large drusen (>= 125 microns) in the study eye and no large drusen or advanced AMD (choroidal neovascularization (CNV) or geographic atrophy (GA)) in the fellow eye. Group 2 (N=40) is defined as participants with bilateral large drusen (>= 125 microns) with or without retinal pigment epithelial hypo/hyperpigmentary changes. Group 3 (N=40) is defined as participants with large drusen (>= 125 microns) in the study eye and advanced AMD (CNV or GA) in the fellow eye. Group 4 (N=40) is defined as participants with findings of reticular pseudodrusen (RPD) defined as having (1) the presence of reticular inter-lacing patterns on at least one en face imaging method (color photography, autofluorescence or infrared) and (2) confirmation of previously described findings of hyperreflective material located between the retinal pigment epithelium (RPE) and the photoreceptor ellipsoid zone on SD OCT in those areas. Current participants in this study have been graded and categorized into this cohort. Up to 40 diabetic participants will be recruited.

Design: This is a single center, exploratory, observational, longitudinal evaluation of dark adaptation response in AMD participants over five years and long-term evaluation of dark adaptometry (DA) change as a predictor for AMD progression and visual acuity (VA) loss.

Outcome Measures: The primary outcome is to determine mean change, including the distribution of change, in dark adaptation response between baseline and months 12 and 24 for Groups 0, 1, 2, 3 and 4. The secondary outcomes for each of the five groups are to determine mean change in dark adaptation response from baseline at months 3, 6, 18, 36, 48 and 60 and to determine mean change in best-corrected visual acuity (BCVA) of the study eye from baseline at months 3, 6, 12, 18, 24, 36, 48 and 60. Exploratory outcomes for each of the five groups are to correlate mean BCVA of the study eye with mean dark adaptation response at baseline and months 3, 6, 12, 18, 24, 36, 48 and 60 and to correlate AMD severity, including grading by an external Reading Center, with dark adaptation response at baseline and months 3, 6, 12, 18, 24, 36, 48 and 60. Images from all visits may be sent to the Reading Center; however, only the baseline and annual visits are required to be graded. This study will also analyze renal function in AMD participants. Additionally, exploratory analysis of the small sample of diabetic participants will also be performed.

Outcome measures for the genetic testing and RNA sequencing performed on participants co-enrolled in the Biobank protocol (12-EI-0042) include the interaction of key parameters of phenotype (such as visual acuity, dark adaptation, and retinal features on ocular imaging) with genetic variants and other biomarkers identified from biospecimens, and the characterization of new experimental models of eye health and disease.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants will be eligible if the following inclusion criteria are met:

* Participant is able to understand and sign the protocol s informed consent document.
* Participant is able to complete and comply with study assessments for the full duration of the study.
* Participant is >= 50 years of age.
* Participant has a BCVA score of >= 20/100 (Snellen equivalent) in study eye.
* Participant qualifies for one of the following groups based on AMD grading as defined below.

  * Group 0: Participant without AMD defined as no large drusen or advanced AMD in either eye;
  * Group 1: Participant has at least one large drusen (>= 125 microns) in the study eye and no large drusen or advanced AMD in the fellow eye;
  * Group 2: Participant has bilateral large drusen (>= 125 microns) with or without retinal pigment epithelial hypo/hyperpigmentary changes;
  * Group 3: Participant has at least one large drusen (>= 125 microns) in the study eye and advanced AMD in the fellow eye.
  * Group 4: Participant has reticular pseudodrusen in the study eye defined as having (1) the presence of RPD on at least one en face imaging method (color photography, autofluorescence or infrared) and (2) confirmation of previously described findings of hyperreflective material located between the RPE and the photoreceptor ellipsoid zone on SD OCT in those areas.

EXCLUSION CRITERIA:

Participants who meet any of the following criteria will be excluded from this study:

* Participant has advanced AMD in the study eye at the baseline visit.
* Participant has other active ocular or macular diseases (e.g., diabetic macular edema, retinal vein occlusion, Stargardt's disease or cone-rod dystrophy) or other known ocular disorders that have caused a visual field deficit (e.g., glaucoma with known visual field defect) in the study eye.
* Participant has a fixation deficit in the study eye that would prevent the participant from performing the AdaptDxTM dark adaptation protocol.
* Participant has a medical condition that the investigator feels would prevent the participant from complying with or being able to complete the study assessments.
* Participant had cataract surgery in the study eye within three months prior to enrollment.
* Participant has an oral intake of high doses of vitamin A palmitate supplement (>= 10,000 international units (IU) per day).
* Participant has or had hepatitis or liver disease. Abnormally low vitamin A can alter dark adaptation and chronic liver disease has been associated with low vitamin A.
* Participant has a history of vitamin A deficiency.
* Participant is an NEI employee or subordinate or co-worker of an investigator.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two hundred forty participants (240) will be initially accrued; however, up to 280 participants who meet the eligibility criteria may be enrolled. In the event that a participant withdraws from the study prior to month 12, an additional participant will be accrued. A maximum of 40 non-diabetic participants per group will be accrued in order to obtain 200 non-diabetic participants for the primary outcome analysis. Every effort will be made to ensure 40 non-diabetic participants per group are accrued. Additionally, a maximum of 40 diabetic participants will be accrued across all groups for the exploratory outcome analysis.
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2011-05-16 (Actual)

PRIMARY OUTCOMES:
The primary outcome is to determine mean change, including the distribution of change, in dark adaptation response between baseline and months 12 and 24 for Groups 0 - 4. | Month 12 and Month 24
  mean change, including the distribution of change, in dark adaptation response

SECONDARY OUTCOMES:
To determine mean change in dark adaptation response from baseline at months 3, 6, 18, 36, 48 and 60 . | Months 3, 6, 18, 36, 48 and 60
  mean change in DA response from baseline
To determine mean BCVA of the study eye from baseline at months 3, 6, 12, 18, 24, 36, 48 and 60. | Months 3, 6, 12, 18, 24, 36, 48 and 60
  mean BCVA of study eye from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Emily Y Chew, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ferris FL 3rd, Fine SL, Hyman L. Age-related macular degeneration and blindness due to neovascular maculopathy. Arch Ophthalmol. 1984 Nov;102(11):1640-2. doi: 10.1001/archopht.1984.01040031330019. PMID 6208888
- [Background] Friedman DS, O'Colmain BJ, Munoz B, Tomany SC, McCarty C, de Jong PT, Nemesure B, Mitchell P, Kempen J; Eye Diseases Prevalence Research Group. Prevalence of age-related macular degeneration in the United States. Arch Ophthalmol. 2004 Apr;122(4):564-72. doi: 10.1001/archopht.122.4.564. PMID 15078675
- [Background] Scilley K, Jackson GR, Cideciyan AV, Maguire MG, Jacobson SG, Owsley C. Early age-related maculopathy and self-reported visual difficulty in daily life. Ophthalmology. 2002 Jul;109(7):1235-42. doi: 10.1016/s0161-6420(02)01060-6. PMID 12093644
- [Background] Grune T, Lietz G, Palou A, Ross AC, Stahl W, Tang G, Thurnham D, Yin SA, Biesalski HK. Beta-carotene is an important vitamin A source for humans. J Nutr. 2010 Dec;140(12):2268S-2285S. doi: 10.3945/jn.109.119024. Epub 2010 Oct 27. PMID 20980645
- [Derived] Duic C, Pfau K, Keenan TDL, Wiley H, Thavikulwat A, Chew EY, Cukras C. Hyperreflective Foci in Age-Related Macular Degeneration are Associated with Disease Severity and Functional Impairment. Ophthalmol Retina. 2023 Apr;7(4):307-317. doi: 10.1016/j.oret.2022.11.006. Epub 2022 Nov 17. PMID 36403926
- [Derived] Hess K, de Silva T, Grisso P, Wiley H, Thavikulwat AT, Keenan TDL, Chew EY, Cukras CA. Evaluation of Cone- and Rod-Mediated Parameters in Dark Adaptation Testing as Outcome Measures in Age-Related Macular Degeneration. Ophthalmol Retina. 2022 Dec;6(12):1173-1184. doi: 10.1016/j.oret.2022.05.018. Epub 2022 May 26. PMID 35643387
- [Derived] Yazdanie M, Alvarez J, Agron E, Wong WT, Wiley HE, Ferris FL 3rd, Chew EY, Cukras C. Decreased Visual Function Scores on a Low Luminance Questionnaire Is Associated with Impaired Dark Adaptation. Ophthalmology. 2017 Sep;124(9):1332-1339. doi: 10.1016/j.ophtha.2017.05.005. Epub 2017 Jun 8. PMID 28602520
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-EI-0147.html